CLINICAL TRIAL: NCT04850534
Title: Evaluation and Prognostic Indications of Systemic Inflammation in Liver Cirrhosis Patients
Brief Title: Systemic Inflammation in Liver Cirrhosis
Acronym: SILC
Status: Completed | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Jinlai Liu, Clinical Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SILC
Record Dates: First submitted 2021-04-18; First posted 2021-04-20 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Systemic inflammation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EGD+NSBB: Patients receiving both endoscopic therapy and non-selective beta-blockers for treating high-risk esophagogastric varices
- EGD: Patients receiving mono endoscopic therapy for treating high-risk esophagogastric varices

SUMMARY:
Investigate systemic inflammation in liver cirrhosis patients

ELIGIBILITY:
Inclusion Criteria:

1. Decompensated liver cirrhosis, with endoscopy-verified high-risk esophagogastric varices;
2. Adult patients aged 18-75 years;
3. Willing to anticipate and informed consent form obtained

Exclusion Criteria:

1. History of prior radio-interventional therapy (TIPS or BRTO), liver transplantation, splenectomy, or hepatectomy;
2. Non-sinusoidal cirrhosis (e.g. vascular cirrhosis);
3. Coexistence with advanced hepatocellular carcinoma or other malignancies;
4. Coexistence with severe systemic diseases and less than 3 months of expected survival time;
5. Acute infection within 4 weeks before recruitment;
6. Antibiotic use within 4 weeks before recruitment;
7. Initial antiviral therapy for HBV or HCV within 4 weeks before recruitment;
8. Pregnant or lactating women;
9. Patients resistant to long-term follow-up

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of liver cirrhosis with high-risk bleeding esophaogastric varices
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Upper Gastrointestinal Bleeding | One Year
  Overt upper GI bleeding due to esophagogastric varices, ulcers and other causes; Identified by clinical manifestations, lab tests and endoscopy and measured by number/proportion of patients
Death | One Year
  Deaths caused by variceal bleeding, hepatocellular carcinoma, liver failure, etc

SECONDARY OUTCOMES:
New or worsening acute decompensation event other than upper GI bleeding | One Year
  Ascites, Hepatic encephalopathy, systemic infection, spontaneous bacterial peritonitis, hepatorenal syndrome, etc Identified by clinical manifestations, lab tests and images according to renown practice guidelines and measured by number/proportion of patients
Liver transplantation/ Transfer to other non-endoscopic therapies | One Year
  Undergo liver transplantation, or transferred to surgical, radio-interventional, or other non-endoscopic therapies; Measured by number/proportion of patients

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wu, Ph.D, Principal Investigator — Department of Gastroenterology, Third Affiliated Hospital of Sun Yar-sen University
Locations (1):
- Department of Cardiology, the Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided